CLINICAL TRIAL: NCT06247605
Title: Phase III Clinical Study of AL8326 Tablets in Patients With Advanced or Recurrent Small Cell Lung Cancer After at Least Prior Second-line Treatment
Brief Title: A Phase IIII Study of AL8326 in Small Cell Lung Cancer
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Advenchen Laboratories Nanjing Ltd. (Industry)
Responsible Party: Sponsor
Organization: Advenchen Laboratories, LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AL8326-GB-010
Record Dates: First submitted 2023-10-09; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Small Cell Lung Carcinoma
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: To maintain study blinding, until the study is completed, it should be Ensure that blinded staff and associated with this trial may not see the random table and treatment group assignments.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- active group（AL8326） (Experimental): Oral AL8326 (28-day cycle, once daily) until confirmation of disease progression, intolerable toxicity or death, voluntary withdrawal from the study, for a total of no more than 12 months (approximately 13 cycles).
  Interventions: Drug: AL8326 tablets
- Control group（Placebo) (Placebo Comparator): Oral placebo (28-day cycle, once daily) until confirmation of disease progression, intolerable toxicity or death, voluntary withdrawal from the study, for a total of no more than 12 months (approximately 13 cycles).
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: AL8326 tablets — 10mg/tablet, Oral administration, once daily.
  Other Names: AL8326
  Arms: active group（AL8326）
Drug: placebo — Oral administration, once daily.
  Arms: Control group（Placebo)

SUMMARY:
This is a multicenter, randomized, double-blind, placebo-controlled, phase III study to evaluate the efficacy and safety of AL8326 tablets in small cell lung cancer (SCLC) patients with disease progression or recurrence after receiving at least second-line treatment regimens.

DETAILED DESCRIPTION:
There are 2 treatment groups in this trial, and the study population, sample size and basic design of each group are:

Patients with pathologically confirmed small cell lung cancer at baseline and need = or >3rd line treatment : the sample size was expected to be 243 cases, 162 in the active group and 81 in the control group.

Subjects will be randomized in a 2:1 ratio under double-blind conditions into two groups, with the active group receiving the trial drug AL8326 tablets and the control group receiving placebo. AL8326 tablets and placebo are administered as follows: oral administration, once daily for 28 days per cycle until intolerable toxicity or established disease progression or death or voluntary withdrawal or up to 12 months ( approximately 13 cycles) of treatment. Subjects will have a final visit, followed by a long-term follow-up period, and the tumor disease status will be determined according to RECIST 1.1.

ELIGIBILITY:
Inclusion Criteria:

1. All subjects or legal representatives must sign the informed consent form approved by the Ethics Committee in writing prior to the start of any screening procedures;
2. Age ≥ 18 years, male or female;
3. Histologically or cytologically confirmed small cell lung cancer patients who have recurrent or advanced disease after at least two lines of systemic regimen (including first-line platinum-based therapy, second-line monotherapy or other therapies *);
4. At least one measurable tumor lesion according to RECIST 1.1 **;
5. Expected survival time of at least 12 weeks;
6. ECOG (PS) score of 0 to 2;
7. Subject has adequate organ and bone marrow function and meets the following laboratory criteria:

   1. Blood routine test (without red blood cell or platelet transfusion or hematopoietic factor drug correction within 14 days before screening): absolute neutrophil count (ANC) ≥ 1.5 × 10^9/L (1500/mm3), platelets ≥ 80 × 10^9/L; hemoglobin ≥ 9.0 g/dL;
   2. Liver function: serum total bilirubin ≤ 1.5 × ULN (upper limit of normal), except for patients with Gilbert 's syndrome (persistent or recurrent hyperbilirubinemia, manifested as unconjugated bilirubin elevation in the absence of hemolysis or pathological evidence of liver); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN for patients without liver metastasis, and ALT and AST ≤ 5 × ULN for patients with liver metastasis;
   3. Renal function: Serum creatinine ≤ 1.5 × ULN and estimated standard cendogenous creatinine clearance rate ≥ 60 ml/min by Cockcroft-Gault formula, Ccr (ml/min) = [(140-age) × body weight (kg)]/[72 × Scr (mg/dl)], calculated for females × 0.85;
   4. Coagulation function: international normalized ratio (INR) ≤ 1.5;
   5. Left ventricular ejection fraction (LVEF) > 50% at screening. 8.1) Female: For female subjects of childbearing potential, they must have a negative serum pregnancy test within 7 days prior to enrollment and agree to use a medically approved method of contraception (condom, sponge, gel, diaphragm, IUD, oral or injectable contraceptive, subcutaneous implant, etc.) during and for 3 months after treatment; they must be non-pregnant and lactating. Female subjects are considered fertile if they are menopausal but have not reached post-menopausal status (menopause of 12 consecutive months or more, with no cause other than menopause) and have not undergone sterilization (removal of ovaries and/or uterus). Their sexual partner agrees to use a medically licensed method of contraception during the subject's treatment and for 3 months after completion; 2) Males: surgical sterilization or agreement to use medically licensed contraception during and for 3 months after the end of treatment; their sexual partners agree to use medically licensed contraception during and for 3 months after the end of the subject's treatment;

9. Capable and willing to comply with protocol requirements during the study and subsequent procedures.

Exclusion Criteria:

1. Known uncontrollable hypersensitivity to AL8326 similar compounds;
2. Having previously used AL8326 tablets;
3. Having or had a history of leptomeningeal disease or leptomeningeal metastases at screening, or confirmed CNS metastases presenting with symptoms of uncontrolled brain metastases, spinal cord compression, or cancerous meningitis within 8 weeks of first dose, except for CNS metastases or spinal cord compression that are clinically stable and do not require corticosteroids and have an interval of greater than 2 weeks between screening and previous treatment (including radiation therapy or surgery);
4. Having or had other neoplasms unless radically treated and with no evidence of recurrence or metastasis within the past 2 years;
5. Having significant gastrointestinal history or current illness, such as inability to swallow, severe peptic ulcer, uncontrollable nausea and vomiting, and clinical difficulty in controlling chronic diarrhea, intestinal obstruction or other chronic gastrointestinal diseases in the past 3 months, which may affect the intake, transport or absorption of drugs as judged by the investigator, or who have previously undergone total gastrectomy;
6. Having other important primary diseases, such as single agent uncontrolled hypertension (systolic blood pressure ≥ 150 mmHg and/or diastolic blood pressure ≥ 95 mmHg), arrhythmia requiring clinical intervention (such as long QT syndrome, QTcF > 470 ms), abnormally prolonged arrhythmia caused by unstable coronary artery disease, decompensated congestive heart failure (New York Heart Association(NYHA) class III or IV) or myocardial infarction, unstable angina pectoris, ascites or pleural effusion with uncontrolled within 6 months before the administration of the investigational product (CTCAE 5.0 ≥ 2), active autoimmune diseases, mental illness, symptomatic or interstitial lung disease requiring treatment, thyroid disease that may seriously affect the trial evaluation;
7. Previously received cytotoxic chemotherapy and/or immunotherapy, and the end of the last dose is at least 4 weeks apart from the first dose of study drug; the end of anti- tumor herb medicine is at least 14 days apart; the end of nitroso or mitomycin was at least 6 weeks apart, and tyrosine kinase inhibitors (TKIs) class molecular targeted drugs were at least 4 weeks apart; the treatment of brain metastases/bone metastases had to be at least 2 weeks apart; and had recovered to ≤ Grade 1 from the toxicity of previous treatment [except for the following: a. alopecia; b. long-term toxicity caused by radiotherapy, which could not be recovered in the judgment of the investigator; c. platinum-induced Grade 2 and the following neurotoxicity such as hearing impairment (according to the Common Terminology Criteria for Adverse Events CTCAE V5.0)];
8. Had arterial thrombosis or severe venous thromboembolic events within 6 months before screening, such as cerebrovascular accident (including transient ischemic attack), deep venous thrombosis and pulmonary embolism;
9. Having imaging findings indicating that the tumor has invaded around important vessels at screening or the tumor is likely to invade important vessels and cause fatal massive hemorrhage during the subsequent study period as judged by the investigator;
10. Uncontrolled infection within 14 days prior to first dose;
11. Screening urine routine showed urine protein ≥ + +, and 24-hour urine protein > 1.0 g;
12. Having active bleeding within 3 months before screening or at high risk of bleeding as judged by the investigator;
13. Been receiving anticoagulants or vitamin K antagonists (e.g., warfarin, heparin, or their analogues) during the screening period [low-dose anticoagulants such as warfarin (no more than 1 mg daily orally), low-dose heparin (no more than 12,000 U daily), or low-dose aspirin (no more than 100 mg daily) were permitted for prophylactic purposes provided INR was ≤ 1.5];
14. Having positive test results for hepatitis C virus (HCV) antibody, treponema pallidum antibody, or human immunodeficiency virus (HIV) antibody, or active hepatitis B (defined as hepatitis B virus HBV DNA ≥ 2000 IU/mL or HBV DNA ≥ 10 ^ 4 copies);
15. Participated in other clinical trials (excluding observational or vitamin studies) within 4 weeks before informed consent;
16. Having received major surgical treatment within 6 weeks prior to screening (patients must be fully recovered and stable before the start of treatment) or serious unhealed wounds, ulcers or fractures at screening;
17. Having a history of organ transplantation or being prepared to undergo organ transplantation;
18. Other reasons that, in the discretion of the investigator, would make participation in this study inappropriate.

Notes:

*1 new line of therapy refers to a change in treatment regimen due to disease progression rather than toxicity or other reasons; after progression on the first treatment, reuse of the same treatment regimen is also a new line of therapy;

** Lesions treated with radiotherapy or locoregional therapy must have radiographic evidence of disease progression to be considered target lesions. If there is only one measurable lesion, the lesion cannot be brain lesion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 243 (Estimated)
Dates: Start 2023-10-26 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | Cycle 1 Day 1 up to 3 years (each cycle is 28 days)
  The time between the date of randomization and the death of the subject from any cause.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | Cycle 1 Day 1 up to 12 months(each cycle is 28 days)
  The period of time between the start of the subject's date of randomization and the first observation of disease progression (based on RECIST 1.1 criteria) or the occurrence of death due to any cause (the earlier of the two occurrences).
Objective remission rate (ORR) | 12 months
  Proportion of subjects achieving CR and PR according to RECIST 1.1.
Duration of remission (DOR) | 12 months
  Time from the start of the first assessment of the tumor as CR or PR to the first assessment of PD or death from any cause.
Disease Control Rate (DCR) | 12 months
  Proportion of subjects achieving CR, PR, and SD.
Adverse Events (AEs) | Cycle 1 Day 1 up to 12 months(each cycle is 28 days)
  According to CTCAE V5.0, AES and abnormal indicators of laboratory tests need to be reported according to treatment group, category and worst grade.
Plasma Concentration | Cycle 1 Day 1，Cycle 2 Day1（±3days），Cycle 4 Day 14（±3days）(each cycle is 28 days)
  Sparse PK samples (plasma concentration time data) of all subjects treated with study drug (AL8326 tablets / placebo) were collected for population pharmacokinetic analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Cheng, Principal Investigator — Jilin Provincial Tumor Hospital
Locations (1):
- JILIN Cancer Hospital, Changchun, Jilin, China